CLINICAL TRIAL: NCT05113186
Title: Lenvatinib in Neo-adjuvant and Adjuvant Therapy for Poor-prognosis BCLC A HepatoCellular Carcinoma Treated by Percutaneous Ablation Procedure in a Curative Intent: Multicentre Pilot Therapeutic Trial
Brief Title: Neoadjuvant and Adjuvant Lenvatinib in HCC Patients Treated by Percutaneous Ablative
Acronym: LENVABLA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP201185
Record Dates: First submitted 2021-07-31; First posted 2021-11-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Lenvatinib; Adjuvant; Neoadjuvant; curative intent; percutaneous ablative
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: a pilot interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant and adjuvant therapy with lenvatinib (Experimental): * Neoadjuvant therapy with lenvatinib to complete a 3-week course, stopping 1 week before the planned date of PA procedure
  * Adjuvant therapy with lenvatinib for 3 months starting after the PA evaluation (± 14 days) The daily dose of lenvatinib will be 12 mg (≥60 kg) or 8 mg (<60 kg). Lenvatinib will be taken within 2 hours after a light meal, preferably in the morning.
  Interventions: Drug: Lenvatinib Pill

INTERVENTIONS:
Drug: Lenvatinib Pill — The design of study is summarized as follows:
  * Neoadjuvant phase with lenvatinib for 21 days (rationale: compromise between expected benefit and acceptable tolerance without compromising ablation procedure)
  * PA of HCC in a curative intent (radiofrequency, microwave or electroporation)
  * Adjuvant phase with lenvatinib for 3 months (rationale: compromise between expected benefit and acceptable tolerance without compromising ablation procedure)
  Other Names: percutaneous ablative procedure

SUMMARY:
Percutaneous ablation (PA) is the only non-surgical curative treatment of hepatocellular carcinoma (HCC). Due to its excellent tolerance, particularly in patients with portal hypertension or bearing comorbidities, it now represents in France nearly 70% of the first-line curative treatment of "in Milan" tumours. For HCC less than 3 cm, ideal indication for percutaneous ablations, results of monopolar radiofrequency ablation (mRFA), are excellent with only 5% of reported non-tumoral control after a first procedure. In addition to mRFA the arsenal of ablations has grown considerably with the emergence of new techniques which allow the expansion of indications for PA, especially in patients with poor prognostic tumors or relatively advanced beyond the Milan criteria. In this setting, multibipolar mode using no touch technique (mbpRFAnt) increases the tumour volume than can be ablated, allowing the removal of large tumors> 5 cm. Inadequate tumour control is then de facto greater in these situations, around 20%. Difficult-to-access tumors can furthermore be treated by percutaneous irreversible electrotroporation (IRE).

Despite a tumor burden accessible for curative ablation, a phenotype of "aggressive" HCC characterized by high rates of local recurrences is yet to be defined. Up to now, several characteristics might define this subtype with a poor-prognosis and include 1) high serum alpha-foetoprotein (AFP) levels, 2) radiological infiltrative form, and 3) histological macrotrabecular subtype. Based on these characteristics, median recurrence-free survival of these patients is usually below 10 months.

High serum AFP level is a well-known predictor of HCC recurrence following curative procedure. In patients treated by percutaneous ablation, regardless of the technique used and irrespective of tumor burden, high baseline serum AFP level has tenaciously been reported as an independent predictor or recurrence..

More recently, the radiological description of infiltrative HCC (as opposed to mass-forming) has been identified as an aggressive from of HCC with a poor prognosis even when eligible for ablation. This aspect is often associated with infra-clinical invasion of the portal veins (PV), leading to poor prognosis. Finally, a "massive macrotrabecular" (MTM) histological subtype of HCC associated with specific molecular features has recently been described. This MTM-HCC subtype, reliably observed in 12% of patients eligible for curative treatment, represents an aggressive form of HCC is an independent predictor of early and overall recurrence following PA, which is retained even after patient stratification according to common clinical, biological, and pathological features of aggressiveness.

The idea of optimizing HCC curative treatments using adjuvant biotherapy, particularly in patients with poor-prognosis tumors in curative intent, is particularly attractive. One trial in adjuvant setting was conducted, the STORM trial, that tested the benefit of sorafenib in curative intent of in Milan HCC. This negative trial included patients within Milan HCC, with an expected low rate of recurrence with only few patients treated by PA.

Lenvatinib is a multikinase inhibitor which has been recently approved as firs-line therapy for advanced HCC. The investigators assume that lenvatinib could have also a synergistic local action with PA in two ways. First, given as neoadjuvant regimen, lenvatinib by reducing tumor and liver perfusion could decrease the global heat sink effect associated with loco-regional blood microcirculation during PA. Second, by carrying on in adjuvant treatment, lenvatinib could decrease the magnitude of non-specific inflammatory angiogenesis around the treatment zone, therefore reducing the risk of locoregional (intrasegmental) cells tumor spreading or promotion.

Given the dismall prognosis of the aforementioned poor-prognosis HCC eligible for PA with an overall median recurrence-free survival below 10 months, the investigators hypothesis is that addition of Lenvatinib as neo- and adjuvant therapy might increase tumour control in these difficult-to-treat patients. Patients combining either high serum AFP levels, infiltrative form or MTM-HCC histological subtype represent 30% of BCLC A stage HCC patients in expert centers, and are the ideal candidates for such trials.

Therefore, the first aim of this proposal is to assess the benefit of lenvatinib in neo- and adjuvant setting combined with curative percutaneous ablation for BCLC A HCC patients considered at high risk of local recurrence (high AFP or infiltrative form or macrotrabecular massive subtype).

DETAILED DESCRIPTION:
Multicenter, 20 hepatology or hepatoGastroenterology and radiology departments in 13 French hospitals (inclusion of patients in 12 centers).

A pilot interventional, prospective, multicenter study.

The design of study is summarized as follows:

* Neoadjuvant phase with lenvatinib for 21 days (rationale: compromise between expected benefit and acceptable tolerance without compromising ablation procedure)
* PA of HCC in a curative intent (radiofrequency, microwave or electroporation)
* Adjuvant phase with lenvatinib for 3 months (rationale: compromise between expected benefit and acceptable tolerance without compromising ablation procedure) Lenvatinib doses will be adapted according to SmPC.

Constitution of a biobank with :

* paraffin and frozen tumoral and non tumoral biopsy sampled at before and after one month of neoadjuvant lenvatinib (second biopsies at the time of the PA procedure)
* Serum, plasma samples before the neoadjuvant lenvatinib, before PA procedure, at 1,3 months of the adjuvant lenvatinib and at month 6.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years
* Histological or radiological diagnosis of HCC, whether new or recurrent following a prior curative therapeutic management > 6 months.
* Barcelona Clinical Liver Cancer (BCLC) stage Category A
* Comprising at least one of the following the following characteristics:
* Single tumour>3 cm≤ 5cm or
* Multiple tumours (max 3 lesions ≤ 3cm) or
* Single tumour between 2 and 3 cm with at least one of the following characteristic:

  * Serum AFP>100 ng/mL
  * Infiltrative form
  * Macro-trabecular subtype (if applicable)
* Patients with HCC amenable for PA as assessed by multidisciplinary board
* At least one uni-dimensional measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to modified RECIST for HCC
* Absence of any portal vein thrombosis
* Liver function status Child-Pugh Class A
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Adequate bone marrow, liver and renal function as assessed by the following laboratory tests:

  * Hemoglobin > 8.5 g/dL
  * Absolute neutrophil count ≥ 1500/mm3 (≥ 1200/mm3 for black/African, American)
  * Platelet count ≥ 60,000/ mm3
  * Total bilirubin ≤ 2 mg/dL
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN)
  * Serum creatinine ≤ 1.5 x ULN
  * Prothrombine time-international normalized ratio (PT-INR) < 2.3 and PTT < 1.5
  * Glomerular Filtration Rate (GFR) ≥ 30 mL/min/1.73 m2
* Life expectancy ≥ 3 months
* Women of childbearing potential (WOCBP) need to accept one effective method of contraception until 1 month after the last lenvatinib intake and avoid pregnancy
* Patients who are sexually active with WOCBP partners need to accept one effective method of contraception until 1 month after lenvatinib intake and men must agree to use adequate contraception
* Patients affiliated to a Social Security System
* Written informed consent signed
* Patient under guardianship or curatorship*
* Satisfactory nutritional status (BMI>18 kg/m² for patients under 70 years old, or ≥21 kg/m² for the patients over 70 years old)
* Patient under guardianship or curatorship*

Exclusion Criteria:

* Patients with recurrence of HCC occurring less than six months after a curative treatment regarded as successful
* BCLC stage >A (1 single lesion >5cm or more than 3 lesions ore multifocal HCC >3cm or vascular invasion or extra-hepatic spread)
* Patients with contraindications to PA

  * Pacemakers or patients who have a history of cardiac arrhythmias or irregular heartbeats (in case of electroporation procedure)
  * Ascites
  * Coagulopathy
  * Ongoing bacterial infection
* Patients with contraindication to contrast medium intravenous injection either gadolinium or iodinate
* Prior liver transplantation
* Prior systemic treatment for HCC (chemotherapy, any other TKI, immunotherapy)
* Patients with large esophageal varices at risk of bleeding that are not being treated with conventional medical intervention
* Past or concurrent history of neoplasm other than HCC, except for in situ carcinoma of the cervix uteri and/or non-melanoma skin cancer and superficial bladder tumours. Any cancer curatively treated > 3 years prior to study entry is permitted
* Major surgical procedure or significant traumatic injury within 28 days before enrolment
* Congestive heart failure New York Heart Association (NYHA) ≥ class 2
* Unstable angina or myocardial infarction within the past 6 months before enrolment
* Uncontrolled blood pressure to systolic BP >140mmHg or diastolic BP >90 mmHg in spite of an optimized regimen of antihypertensive medication.
* Patients with phaeochromocytoma
* Refractory ascites according to EASL guidelines definition (ascites that cannot be mobilized or the early recurrence of which cannot be prevented because of a lack of response to sodium restriction and diuretic treatment)
* Persistent proteinuria of NCI-CTCAE version 4.0 ≥ Grade 3
* Ongoing infection > Grade 2 according to NCI-CTCAE version 4.0. Hepatitis B is allowed if no active replication is present (below 100 IU/mL). Hepatitis C is allowed if no antiviral treatment is required
* Clinically significant bleeding NCI-CTCAE version 4.0 ≥ Grade 3 within 30 days before enrolment
* Any psychological, familial, sociological, geographical or illness or medical condition that could jeopardize the safety of the patient and/or his compliance with the study protocol and follow-up procedure
* Non-healing wound, ulcer or bone fracture
* Known hypersensitivity to the study drug or excipients in the formulation
* Any malabsorption condition
* Breast feeding
* Pregnancy
* Patient unable to swallow oral medication

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
One-year local recurrence-free survival | At one year
  Recurrence rate local will be assessed using imaging techniques as recommended by international guidelines (3-months US and MRI during two years). Patients who will meet primary endpoint will be alive 1 year afterPA procedure without evidence of local recurrence on 3-months US/MRI evaluations.

SECONDARY OUTCOMES:
Per nodule assessment of early response (one month) after PA | At one month after a single procedure of PA
  Evaluation performed by MRI : Assessment of complete response versus incomplete response (persistence of active tumour).
  Evaluation performed by MRI
Per nodule assessment of local recurrence | During 2 years following PA procedure
  Evaluation performed by MRI

OTHER OUTCOMES:
Per nodule assessment of intra segmental distant recurrence | During 2 years following PA procedure
  Evaluation performed by MRI
Per nodule assessment of extra segmental distant recurrence | During 2 years following PA procedure
  Evaluation performed by MRI
Assessment of overall recurrence-free survival at 1 and 2 years | At 1 year and 2 years following PA procedure
  patients will meet this endpoint if they are alive with or without HCC recurrenceat 1and 2 years after PA procedure. Causes and date of death will be specified when applicable during this timeframe.
Evaluation of the safety of lenvatinib administered as neo and adjuvant therapy | During 2 years of follow up
  Adverse events related : fatigue, arterial hypertension, hand-foot skin syndrome to Lenvatinib will be monitored according to manufacturer guidelines and recommendation
Assessment of tumour architecture and cytology : Histological outcome measures | from inclusion to Percutaneous Ablation procedure; assessed up to 30 days
  Absence of tumour cells (binary scale :0/1)
Assessment of tumour architecture and cytology :Histological outcome measures | from inclusion to Percutaneous Ablation procedure; assessed up to 30 days
  Assessment of intra and extra tumoral inflammatory infiltrate (semi quantitative scale: 0=non, 1=mild, 2=intense)
Assessment of tumour architecture and cytology :Genomics | from inclusion to Percutaneous Ablation procedure; assessed up to 30 days
  change in gene expression following sequential whole exome sequencing (binary scale 0/1 with clustering analyses)
Compliance to lenvatinib treatment :Number of returned capsules | during 3-weeks for the neodjuvant lenvatinib and 3 months starting after the PA evaluation
  Accounting for treatment returns. checking respect of scheduled lenvatinib administered
Absence of tumour cells (binary scale: 0/1) | At inclusion, and at the time of the PA procedure
  Consittution of a sequential biobank comprising liver tissue : histological outcome
Assessment of intra and extra tumoral inflammatory infiltrate (semi quantitative scale: 0=non, 1=mild, 2=intense)outcome | At inclusion, and at the time of the PA procedure
  Consittution of a sequential biobank comprising liver tissue : histological
Consittution of a sequential biobank comprising liver tissue : Genomics | At inclusion, and at the time of the PA procedure
  change in gene expression following sequential whole exome sequencing (binary scale 0/1 with clustering analyses)
Consittution of a sequential biobank comprising peripheral samples (serum, plasma) | At inclusion,at Percutaneous Ablation ; at 1, 3 and 6 months after PA
  Changes in PIGF (UI/mL), VEGF-A (UI/mL), VEGF-C (UI/mL), sVEGFR2 (UI/mL), sVEGFR3 (UI/mL), MET (UI/mL), sKIT (UI/mL), Ang2 (UI/mL), AFP (UI/mL), PIVKA (UI/mL) (changes expressed by median comparison)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre NAHON, MD-PhD, Principal Investigator — APHP-Hôpital Jean Verdier
Locations (1):
- NAHON, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nault JC, Sutter O, Nahon P, Ganne-Carrie N, Seror O. Percutaneous treatment of hepatocellular carcinoma: State of the art and innovations. J Hepatol. 2018 Apr;68(4):783-797. doi: 10.1016/j.jhep.2017.10.004. Epub 2017 Oct 13. PMID 29031662
- [Background] N'Kontchou G, Nault JC, Sutter O, Bourcier V, Coderc E, Grando V, Nahon P, Ganne-Carrie N, Diallo A, Sellier N, Seror O. Multibipolar Radiofrequency Ablation for the Treatment of Mass-Forming and Infiltrative Hepatocellular Carcinomas > 5 cm: Long-Term Results. Liver Cancer. 2019 May;8(3):172-185. doi: 10.1159/000489319. Epub 2018 Jun 28. PMID 31192154
- [Background] Sutter O, Calvo J, N'Kontchou G, Nault JC, Ourabia R, Nahon P, Ganne-Carrie N, Bourcier V, Zentar N, Bouhafs F, Sellier N, Diallo A, Seror O. Safety and Efficacy of Irreversible Electroporation for the Treatment of Hepatocellular Carcinoma Not Amenable to Thermal Ablation Techniques: A Retrospective Single-Center Case Series. Radiology. 2017 Sep;284(3):877-886. doi: 10.1148/radiol.2017161413. Epub 2017 Apr 28. PMID 28453431
- [Background] Ziol M, Pote N, Amaddeo G, Laurent A, Nault JC, Oberti F, Costentin C, Michalak S, Bouattour M, Francoz C, Pageaux GP, Ramos J, Decaens T, Luciani A, Guiu B, Vilgrain V, Aube C, Derman J, Charpy C, Zucman-Rossi J, Barget N, Seror O, Ganne-Carrie N, Paradis V, Calderaro J. Macrotrabecular-massive hepatocellular carcinoma: A distinctive histological subtype with clinical relevance. Hepatology. 2018 Jul;68(1):103-112. doi: 10.1002/hep.29762. Epub 2018 May 9. PMID 29281854
- [Background] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850